CLINICAL TRIAL: NCT01725646
Title: A Randomized, Double-blinded, Placebo-controlled Study to Assess the Efficacy and Safety of Omacor® in Taiwanese Hypertriglyceridemic Patients
Brief Title: An Efficacy and Safety Study of Omacor® in Taiwanese Hypertriglyceridemic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Excelsior (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OM3-99001
Record Dates: First submitted 2012-10-29; First posted 2012-11-14 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia, omega-3-acid ethyl ester
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omacor® 4 g (Active Comparator): Subjects in this group will take 4 g of Omacor® everyday.
  Interventions: Drug: Omacor®
- Omacor® 2 g (Active Comparator): Subjects in this group will take 2 g of Omacor® and 2 g of placebo everyday.
  Interventions: Drug: Omacor®
- Placebo (Placebo Comparator): Subjects in this group will take 4 g of placebo everyday.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omacor® — Subjects in 4 g and 2 g Omacor® will take this drug
  Other Names: Omega-3-acid ethyl ester 90
  Arms: Omacor® 2 g; Omacor® 4 g
Drug: Placebo — Subjects in placebo group will take this drug
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
1. Evaluation of the efficacy of Omacor® in Taiwanese hypertriglyceridemia patients
2. Evaluation of the safety of Omacor® in Taiwanese hypertriglyceridemia patients

DETAILED DESCRIPTION:
The primary end point is to evaluate the efficacy and safety of Omacor in Taiwanese hypertriglyceridemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has fasting serum TG ≥ 200 mg/dL but no more than 1000 mg/dL

Exclusion Criteria:

* Patients had a history of pancreatitis or considered to be at risk of developing pancreatitis
* Patient had history of a severe cardiovascular event or a revascularization procedure within 6 months prior to randomization

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Triglycerides from baseline | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Den Tseng, M.D., PhD., Principal Investigator — NTUH
Locations (4):
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Veterans General Hospital, Taipei, Taiwan